CLINICAL TRIAL: NCT02993224
Title: Open-label, Multicenter, Single Arm, Phase II Study Assessing Treatment Patient Preference for New Deferasirox Formulation (Film-coated Tablet) Compared to the Reference Deferasirox Dispersible Tablet Formulation
Brief Title: Open-label, Multicenter Study Assessing Preference for Deferasirox Film-coated Tablet Compared to Dispersible Tablet
Acronym: Jupiter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CICL670FIC05; 2016-002282-61 (EudraCT Number)
Record Dates: First submitted 2016-11-08; First posted 2016-12-15 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Transfusion-dependent Thalassemia; Non-transfusion-dependent Thalassemia
Keywords: thalassemia; TDT; transfusion-dependent; non-transfusion-dependent; NTDT
MeSH Terms: conditions — Thalassemia | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferasirox DT followed by deferasirox FCT (Experimental): Participants were treated with deferasirox DT followed by deferasirox FCT (core phase). Those who entered the extension phase were treated with deferasirox FCT
  Interventions: Drug: Deferasirox dispersable tablet (DT); Drug: Deferasirox film coated tablet (FCT)

INTERVENTIONS:
Drug: Deferasirox dispersable tablet (DT) — Deferasirox DT was provided as 125 mg, 250 mg, 500 mg dispersible tablets for oral use. The strengths provided in an individual country could differ and reflected the strengths available commercially in each country.
  For iron chelation naive participants, the starting dose on Baseline Day 1 was 20 mg/kg/day in TDT and 10 mg/kg/day in NTDT.
  For iron chelation (deferoxamine and/or deferiprone) pre-treated participants, the starting dose was equivalent to the dose of deferoxamine received (for participants pre-treated with deferoxamine) and based on their serum ferritin levels (for participants pre-treated with deferiprone).
  Participants took deferasirox DT once daily for 24 weeks (core phase). The required number of deferasirox DT tablets were to be dispersed with gentle stirring in a glass of water.
Drug: Deferasirox film coated tablet (FCT) — Deferasirox FCT was provided as 90 mg, 180 mg, 360 mg film coated tablets for oral use. The FCT starting dose on Week 25 was 14 mg/kg/day in TDT and 7 mg/kg/day in NTDT.
  Participants took deferasirox FCT once daily for 24 weeks during the core phase and up to 48 weeks during the extension phase. For patients with difficulties in swallowing deferasirox FCT, it was allowed to crush the film-coated tablets and administer the study drug by sprinkling the full dose on soft food (like yogurt or apple puree).

SUMMARY:
Study to evaluate patient preference of deferasirox film-coated tablet (FCT) or deferasirox dispersible tablet (DT) in patient with transfusion - dependent thalassemia or non-transfusion -dependent thalassemia as measured by preference questionnaire at Week 48

DETAILED DESCRIPTION:
This was an open-label, multicenter, single arm, phase II study aimed at collecting data on preference for iron chelation therapy in patients with transfusion-dependent thalassemia (TDT) or non-transfusion-dependent thalassemia (NTDT) throughout a 48 week treatment period. Participants who were either chelator-naïve, or who were previously treated with iron chelators (excluding deferasirox) for at least 6 months continuously, were eligible to participate in this study.

The study was divided into 2 phases:

1. Core Phase:

   * Screening phase which lasted for a maximum of 4 weeks to determine patient eligibility followed by
   * Period 1: Participants were treated with deferasirox DT from Baseline visit Day 1 to Week 24
   * Period 2: Participants were treated with deferasirox FCT from Week 25 to Week 48:

   At the discretion of the investigator, patients could switch from deferasirox DT to deferasirox FCT at any time during Period 1 of the Core phase, and vice versa, from deferasirox FCT to deferasirox DT at any time during Period 2 of the Core phase. Re-switching treatments was not allowed within each period.
2. Extension Phase:

Participants could continue deferasirox FCT formulation as per the judgment of the investigator, through an extension phase for a maximum of 48 weeks months from the last dose of deferasirox FCT received at the end of period 2 in the Core Phase or until one of the end of study criteria defined is met, whichever came first. Participation in the extension phase was optional.

The end of study was defined as the earliest occurrence of one of the following:

* The patient reached Week 96 in the Extension phase.
* Deferasirox FCT was locally reimbursed for this indication (only applicable for the Extension phase)
* Another clinical study or post-trial access program became available that could continue to provide deferasirox FCT in this patient population and all patients ongoing were eligible to be transferred to that clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to any screening procedures were performed, written informed consent/assent must be provided. For pediatric patients, consent was obtained from parent(s) or legal patient's representative. Investigators also obtained assent of patients according to local, regional or national guidelines.
2. Male and female patient aged ≥ 2 years
3. Deferasirox naïve patient or chelated naive patient or treated by other chelators for at least 6 months, such as:

   1. Deferiprone/ DFP
   2. Deferoxamine /DFO
   3. Combination (DFO + DFP)
4. Subject was willing to discontinue current iron chelation therapy at least 5 days prior to study day 1 and for the duration of the study
5. Patients with transfusion-dependent thalassemia (independent of underlying condition) with transfusional iron overload as shown by a serum ferritin level of > 1000 ng/ml at screening and if available, LIC > 3 mg Fe/g dw within 6 months prior to screening
6. Patients with non-transfusion-dependent thalassemia with iron overload as shown by a serum ferritin level of ≥ 800 ng/ml at screening and if available, LIC ≥ 5 mg Fe/g dw within 6 months prior to screening

Exclusion Criteria:

1. Creatinine clearance below the contraindication limit in the locally approved prescribing information.
2. Serum creatinine level > 1.5 x ULN (upper limit of normal)
3. AST (SGOT) /ALT (SGPT) > 5 x ULN, unless LIC confirmed as >10 mg Fe/dw within 6 months prior to screening visit.
4. Significant proteinuria as indicated by a urinary protein/creatinine ratio > 0.5 mg/mg in a non-first void urine sample.
5. Patients with significant impaired gastrointestinal (GI) function or GI disease that might significantly alter the absorption of oral deferasirox (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
6. Clinical or laboratory evidence of active Hepatitis B or Hepatitis C (HBsAg in the absence of HBsAb OR HCV Ab positive with HCV RNA positive).
7. Patients with psychiatric or addictive disorders which prevent them from giving their informed consent or undergoing any of the treatment options or patients unwilling or unable to comply with the protocol
8. Patients with a known history of HIV seropositivity (Elisa or Western blot).
9. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
10. Patients participating in another clinical trial or receiving an investigational drug. Patients who have recently completed treatment with an investigational product must have ceased this treatment for at least five times the half-life of the investigational product.
11. History of hypersensitivity to any of the study drug or excipients.
12. Significant medical condition interfering with the ability to partake in this study (e.g. systemic uncontrolled hypertension, unstable cardiac disease not controlled by standard medical therapy, systemic disease (cardiovascular, renal, hepatic, etc.).
13. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using effective methods of contraception during dosing of study treatment
14. Women were considered post-menopausal and not of child bearing potential if they had had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or had had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
15. Sexually active males unless they used a condom during intercourse while taking drug and for 28 days after stopping study medication and should not father a child in this period. A condom was required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Egypt (3):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
  - Novartis Investigative Site, Zagazig
- Novartis Investigative Site, Hazmiyeh, Beyrouth, Lebanon
- Novartis Investigative Site, Rabat, Morocco
- Saudi Arabia (3):
  - Novartis Investigative Site, Al Ahsa, SAU
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Thailand (3):
  - Novartis Investigative Site, Bangkok Noi, Bangkok
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 17 investigative sites in 7 countries
Period: Core Phase - Period 1
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Started | 148
Completed | 140
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3
Period: Core Phase- Period 2
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Started | 140
Completed | 136
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Unwillingness To Comply With Protocol Procedures And Prescribed Study Treatment | 2
Not completed — Allogenic stem cell transplantation | 1
Period: Extension Phase
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Started (Participation in the extension phase was optional) | 116
Completed | 80
Not Completed | 36
Not completed — Unwillingness To Comply With Protocol Procedures And Prescribed Study Treatment | 1
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Deferasirox FCT locally reimbursed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.32 (13.824)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian (Indian subcontinent) | 5
  Other | 143

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Preferring Deferasirox FCT or DT at Week 48 Based on Preference Questionnaire (Item 2)
Description: Number of participants preferring deferasirox FCT or DT as measured by preference questionnaire (item 2) at Week 48. The preference questionnaire was a 3-item questionnaire. At Week 48, the second item of the preference questionnaire asked the patients (or parents of young patients from 2 to 9 years old) which medicine did the patient "like best": "Tablet to dissolve in liquid" (=deferasirox DT), "Film coated tablet" (=deferasirox FCT), "Sprinkle powder on food" (=deferasirox FCT) and "I don't know" (=none of the above). The number of participants who selected each response option for item 2 was assessed. The analysis was performed for participants who answered the item 2 of the preference questionnaire.
Time Frame: Week 48
Population: Full Analysis Set (FAS): Participants to whom study treatment was assigned and who received at least one dose of each study treatment (DT and FCT). Only participants with available data for this outcome measure were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 134
Participants
  Preference for deferasirox DT | 10
  Preference for deferasirox FCT | 121
  Preference for none of the above | 3
Statistical Analysis 1: Comparison: Deferasirox DT Followed by Deferasirox FCT; Preference for deferasirox DT vs deferasirox FCT; Test type: Superiority; p < .0001, McNemar; Difference of proportion = 0.83, 95% CI 2-sided [0.75 to 0.89]

2. Secondary Outcome: Number of Participants Preferring Deferasirox FCT, Deferasirox DT or Previous Iron Chelation Therapy at Week 28 Based on Preference Questionnaire (Item 2)
Description: Number of participants preferring deferasirox FCT, deferasirox DT or previous iron chelation therapy as measured by preference questionnaire (item 2) at Week 28. The preference questionnaire was a 3-item questionnaire. At Week 28, the second item of this questionnaire asked the patients (or parents of young patients from 2 to 9 years old) which medicine did the patient "like best": "Tablet to dissolve in liquid" (=deferasirox DT), "Film coated tablet (taken once a day)" (=deferasirox FCT), "Sprinkle powder on food" (=deferasirox FCT), "Tablet (taken 3 times a day)" (=previous iron chelation therapy), "Injection" (=previous iron chelation therapy) and "I don't know" (=none of the above). The number of participants who selected each response option for item 2 was assessed. This analysis was performed only for patients who had received iron chelation therapy prior to enrolling in the study and who answered the item 2 of the preference questionnaire.
Time Frame: Week 28
Population: Participants in the FAS [to whom study treatment was assigned and who received at least one dose of each study treatment (DT and FCT)] and who received iron chelation therapy prior to enrolling in the study. Only participants with available data for this outcome measure were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 69
Participants
  Preference for deferasirox DT | 6
  Preference for deferasirox FCT | 60
  Preference for previous iron chelation therapy | 3
  Preference for none of the above | 0
Statistical Analysis 1: Comparison: Deferasirox DT Followed by Deferasirox FCT; Preference of deferasirox FCT vs deferasirox DT; Test type: Superiority; p < 0.0001, McNemar; Difference of proportion = 0.78, 95% CI 2-sided [0.65 to 0.88]
Statistical Analysis 2: Comparison: Deferasirox DT Followed by Deferasirox FCT; Preference for deferasirox FCT vs previous iron chelation therapy; Test type: Superiority; p < 0.0001, McNemar; Difference of proportion = 0.83, 95% CI 2-sided [0.71 to 0.91]

3. Secondary Outcome: Number of Participants Preferring Deferasirox DT or Previous Iron Chelation Therapy at Week 4 and Week 24 Based on Preference Questionnaire (Item 2)
Description: Number of participants preferring deferasirox DT or previous iron chelation therapy as measured by preference questionnaire (item 2) at Week 4 and 24. The preference questionnaire was a 3-item questionnaire. At Week 4 and 24, the second item of the preference questionnaire asked the patients (or parents of young patients from 2 to 9 years old) which medicine did the patient "like best": "Tablet to dissolve in liquid" (=deferasirox DT), "Tablet (taken 3 times a day)" (=previous iron chelation therapy), "Injection" (=previous iron chelation therapy) and "I don't know" (=none of the above). The number of participants who selected each response option for item 2 was assessed. This analysis was performed only for patients who had received iron chelation therapy prior to enrolling in the study and who answered item 2 of the preference questionnaire.
Time Frame: Week 4 and Week 24
Population: Participants in the FAS [to whom study treatment was assigned and who received at least one dose of each study treatment (DT and FCT)] and who received iron chelation therapy prior to enrolling in the study. Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 70
Participants
  Week 4: Preference for deferasirox DT | 57
  Week 4: Preference for previous iron chelation therapy | 11
  Week 4: Preference for none of the above | 2
  Week 24: number analyzed (Participants) | 69
  Week 24: Preference for deferasirox DT | 52
  Week 24: Preference for previous iron chelation therapy | 11
  Week 24: Preference for none of the above | 6
Statistical Analysis 1: Comparison: Deferasirox DT Followed by Deferasirox FCT; Deferasirox DT vs previous iron chelation therapy at Week 4; Test type: Superiority; p < 0.0001, McNemar; Difference of proportion = 0.66, 95% CI 2-sided [0.51 to 0.77]
Statistical Analysis 2: Comparison: Deferasirox DT Followed by Deferasirox FCT; Deferasirox DT vs previous iron chelation therapy at Week 24; Test type: Superiority; p < 0.0001, McNemar; Difference of proportion = 0.59, 95% CI 2-sided [0.44 to 0.72]

4. Secondary Outcome: Number of Participants Selecting Each Reason for Treatment Preference as Assessed by the Preference Questionnaire at Week 28 and Week 48
Description: The preference questionnaire was a 3 item questionnaire. The first item asked the patients (or parents of young patients from 2 to 9 years old) which medicine they were taking. The second item asked which of the medicines did the patient "Like best". Finally, the third item asked the patient why he/she preferred the medicine they chose in the second item. The number of participants who selected each response option for item 3 was assessed. Participants could select multiple reasons for treatment preference at each timepoint.
Time Frame: Week 28 and Week 48
Population: FAS: Participants to whom study treatment was assigned and who received at least one dose of each study treatment (DT and FCT).
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Participants
  Aftertaste (Week 28) | 9
  Can correctly prepare the medicine (Week 28) | 35
  Convenience (it's not a problem to take your medicine) (Week 28) | 109
  Easier to remember to take the medicine (Week 28) | 57
  Gain my personal time with family and friends (Week 28) | 35
  No/ less pain on the injection site (Week 28) | 31
  No/ less side effects (Week 28) | 50
  Number of pills (Week 28) | 46
  Number of times you have to take the medicine (Week 28) | 42
  Other (Week 28) | 5
  Taste (Week 28) | 30
  Aftertaste (Week 48) | 17
  Can correctly prepare the medicine (Week 48) | 48
  Convenience (it's not a problem to take your medicine) (Week 48) | 103
  Easier to remember to take the medicine (Week 48) | 61
  Gain my personal time with family and friends (Week 48) | 36
  No/ less pain on the injection site (Week 48) | 37
  No/ less side effects (Week 48) | 48
  Number of pills (Week 48) | 41
  Number of times you have to take the medicine (Week 48) | 47
  Other (Week 48) | 0
  Taste (Week 48) | 51

5. Secondary Outcome: Percentage of Consumed Tablet Counts During Deferasirox DT and Deferasirox FCT Treatment Periods
Description: The percentage of consumed tablet counts (compliance) was calculated for each treatment period in the core phase: deferasirox DT (period 1) and deferasirox FCT (period 2). Compliance was defined as the total tablet count consumed divided by total tablet count prescribed and multiplied by 100. Total tablet count consumed was calculated as total number of tablets dispensed minus total number of tablets lost/wasted or returned. Total tablet count prescribed was calculated as the number of tablets that the patient should have taken during this period. If a patient did not return the study drug, the compliance was not calculated.
Time Frame: Deferasirox DT: From Baseline up to Week 24. Deferasirox FCT: From Week 25 up to Week 48
Population: FAS: Participants to whom study treatment was assigned and who received at least one dose of each study treatment (DT and FCT). Number analyzed signified number of participants with available data for this outcome measure for each treatment period
Measure: Mean (Standard Deviation); unit: Percentage of tablet counts
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Percentage of tablet counts
  Deferasirox DT (Baseline up to Week 24) | 98.68 (22.373)
  Deferasirox FCT (From Week 25 up to Week 48): number analyzed (Participants) | 138
  Deferasirox FCT (From Week 25 up to Week 48) | 95.07 (15.368)
Statistical Analysis 1: Comparison: Deferasirox DT Followed by Deferasirox FCT; Compliance of deferasirox DT vs deferasirox FCT; Test type: Superiority; p = 0.1191, ANCOVA; Least squares mean = -3.6, 95% CI 2-sided [-8.1 to 0.9], Standard Error of Mean 2.30

6. Secondary Outcome: Change Over Time in Aftertaste Score of Palatability Questionnaire
Description: The palatability questionnaire consisted of 4 items, three items measuring taste and one item measuring aftertaste. The aftertaste item scored on a 5-point response scale with the response option: Very good = 1, Good = 2, Neither good nor bad = 3, Bad = 4, Very bad = 5. This item offered an additional response option of "no aftertaste". The aftertaste score was calculated among participants who had an aftertaste. Higher aftertaste scores indicated a worse aftertaste.
  For participants less than (<) 10 years old, an observer palatability questionnaire was administered. Items and scoring algorithm remained the same as for participants greater than or equal to (≥) 10 years old.
  Change in aftertaste score over time was assessed
Time Frame: Week 4, 24, 28 and 48
Population: FAS: Participants to whom study treatment was assigned and who received at least one dose of each study treatment (DT and FCT). Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Score on a Scale
  From Week 4 to Week 24 in participants treated with deferasirox DT at Week 24: number analyzed (Participants) | 102
  From Week 4 to Week 24 in participants treated with deferasirox DT at Week 24 | -0.1 (0.80)
  From Week 4 to Week 24 in participants treated with deferasirox FCT at Week 24: number analyzed (Participants) | 6
  From Week 4 to Week 24 in participants treated with deferasirox FCT at Week 24 | -0.5 (1.22)
  From Week 24 to Week 28 in participants treated with deferasirox DT at Week 28: number analyzed (Participants) | 0
  From Week 24 to Week 28 in participants treated with deferasirox FCT at Week 28: number analyzed (Participants) | 106
  From Week 24 to Week 28 in participants treated with deferasirox FCT at Week 28 | -0.5 (1.16)
  From Week 24 to Week 48 in participants treated with deferasirox DT at Week 48: number analyzed (Participants) | 0
  From Week 24 to Week 48 in participants treated with deferasirox FCT at Week 48: number analyzed (Participants) | 98
  From Week 24 to Week 48 in participants treated with deferasirox FCT at Week 48 | -0.5 (1.08)

7. Secondary Outcome: Change Over Time in Palatability Score of Palatability Questionnaire
Description: The palatability questionnaire consisted of 4 items, three items measuring taste and one item measuring aftertaste. Among the taste items, first one measured taste on a 5-point response scale. The other two items measured what happened after taking the medicine and how the perceived amount of liquid taken with the medicine was. Responses to these 3 items were combined and converted into a single palatability score using a scoring matrix: each combination of responses on each of 3 items corresponded to a predefined palatability score. E.g. if a participant responded "bad" to item 1, "vomited <30min" to item 2 and "not enough" to item 3, then the palatability score assigned was 0. This score ranged from 0 to 11; higher scores indicated better palatability. For participants <10 years old, an observer palatability questionnaire was administered. Items and scoring algorithm were the same as for participants ≥10 years old. Change in palatability score over time was assessed
Time Frame: Week 4, 24, 28 and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Score on a Scale
  From Week 4 to Week 24- participants treated with deferasirox DT at Week 24: number analyzed (Participants) | 131
  From Week 4 to Week 24- participants treated with deferasirox DT at Week 24 | -0.1 (2.46)
  From Week 4 to Week 24 in participants treated with deferasirox FCT at Week 24: number analyzed (Participants) | 7
  From Week 4 to Week 24 in participants treated with deferasirox FCT at Week 24 | 0.0 (0.00)
  From Week 24 to Week 28 in participants treated with deferasirox DT at Week 28: number analyzed (Participants) | 0
  From Week 24 to Week 28 in participants treated with deferasirox FCT at Week 28: number analyzed (Participants) | 137
  From Week 24 to Week 28 in participants treated with deferasirox FCT at Week 28 | 1.1 (2.77)
  From Week 24 to Week 48 in participants treated with deferasirox DT at Week 48: number analyzed (Participants) | 0
  From Week 24 to Week 48 in participants treated with deferasirox FCT at Week 48: number analyzed (Participants) | 134
  From Week 24 to Week 48 in participants treated with deferasirox FCT at Week 48 | 1.3 (2.54)

8. Secondary Outcome: Change From Baseline in Adherence Domain Score of Modified Satisfaction With Iron Chelation (mSICT) Questionnaire
Description: The mSICT patient reported outcome (PRO) consisted of 15 items that represented 3 domains: Adherence, Preference, and Concerns. The adherence domain score consisted of 6 adherence items, measured using a 5-point response scale. The adherence score was calculated by summing these 6 items, with scores ranging from 6 to 30. Higher scores indicated worse adherence.
  For participants <10 years old, an observer version (ObsRO) was administered. The adherence score remained the same as for participants ≥10 years old.
Time Frame: Baseline (week 2 or, if missing, week 3), week 24, 28 and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Score on a scale
  Week 24- participants ≥ 10 years treated with deferasirox DT (PRO): number analyzed (Participants) | 72
  Week 24- participants ≥ 10 years treated with deferasirox DT (PRO) | -0.3 (3.37)
  Week 24 - participants ≥ 10 years treated with deferasirox FCT (PRO): number analyzed (Participants) | 4
  Week 24 - participants ≥ 10 years treated with deferasirox FCT (PRO) | -1.0 (2.94)
  Week 28 - participants ≥ 10 years treated with deferasirox DT (PRO): number analyzed (Participants) | 0
  Week 28 - participants ≥ 10 years treated with deferasirox FCT (PRO): number analyzed (Participants) | 77
  Week 28 - participants ≥ 10 years treated with deferasirox FCT (PRO) | 0.5 (3.59)
  Week 48 - participants ≥ 10 years treated with deferasirox DT (PRO): number analyzed (Participants) | 0
  Week 48 - participants ≥ 10 years treated with deferasirox FCT (PRO): number analyzed (Participants) | 75
  Week 48 - participants ≥ 10 years treated with deferasirox FCT (PRO) | 0.5 (3.29)
  Week 24 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 56
  Week 24 - participants < 10 years treated with deferasirox DT (ObsRO) | -0.2 (3.35)
  Week 24 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 3
  Week 24 - participants < 10 years treated with deferasirox FCT (ObsRO) | -0.7 (4.16)
  Week 28 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 0
  Week 28 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 58
  Week 28 - participants < 10 years treated with deferasirox FCT (ObsRO) | 0.8 (3.68)
  Week 48 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 0
  Week 48 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 55
  Week 48 - participants < 10 years treated with deferasirox FCT (ObsRO) | 1.1 (3.79)

9. Secondary Outcome: Change From Baseline in Preference Domain Score of Modified Satisfaction With Iron Chelation (mSICT) Questionnaire
Description: The mSICT patient reported outcome (PRO) consisted of 15 items that represented 3 domains: Adherence, Preference, and Concerns.
  The preference/satisfaction domain score consisted of 2 preference/satisfaction items, measured using a 5-point response scale. The preference score was calculated by summing these 2 items, with scores ranging from 2 to 10. Higher scores indicated worse satisfaction.
  For participants < 10 years old, an observer version (ObsRO) was administered. Preference score remained the same as for participants ≥ 10 years old.
Time Frame: Baseline (week 2 or, if missing, week 3), week 24, 28 and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Score on a scale
  Week 24 - participants ≥ 10 treated with deferasirox DT (PRO): number analyzed (Participants) | 72
  Week 24 - participants ≥ 10 treated with deferasirox DT (PRO) | 0.5 (1.21)
  Week 24 - participants ≥ 10 treated with deferasirox FCT (PRO): number analyzed (Participants) | 4
  Week 24 - participants ≥ 10 treated with deferasirox FCT (PRO) | 0.5 (3.70)
  Week 28 - participants ≥ 10 treated with deferasirox DT (PRO): number analyzed (Participants) | 0
  Week 28 - participants ≥ 10 treated with deferasirox FCT (PRO): number analyzed (Participants) | 77
  Week 28 - participants ≥ 10 treated with deferasirox FCT (PRO) | -1.1 (1.83)
  Week 48 - participants ≥ 10 treated with deferasirox DT (PRO): number analyzed (Participants) | 0
  Week 48 - participants ≥ 10 treated with deferasirox FCT (PRO): number analyzed (Participants) | 75
  Week 48 - participants ≥ 10 treated with deferasirox FCT (PRO) | -0.9 (2.02)
  Week 24 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 55
  Week 24 - participants < 10 years treated with deferasirox DT (ObsRO) | 0.0 (1.49)
  Week 24 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 3
  Week 24 - participants < 10 years treated with deferasirox FCT (ObsRO) | 0.0 (1.73)
  Week 28 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 0
  Week 28 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 57
  Week 28 - participants < 10 years treated with deferasirox FCT (ObsRO) | -0.8 (1.74)
  Week 48 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 0
  Week 48 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 54
  Week 48 - participants < 10 years treated with deferasirox FCT (ObsRO) | -0.9 (1.75)

10. Secondary Outcome: Change From Baseline in Concerns Domain Score of Modified Satisfaction With Iron Chelation (mSICT) Questionnaire
Description: The mSICT patient reported outcome (PRO) consisted of 15 items that represented 3 domains: Adherence, Preference, and Concerns.
  The concerns domain score consisted of 3 items to address any concerns or worries with the medication. All 3 items were measured on a 5-point response scale. The concerns score was calculated by summing the 3 items, with scores ranging from 3 to 15. Higher scores indicated fewer concerns. For participants < 10 years old, an observer version (ObsRO) was administered. Concerns score remained the same as for participants ≥ 10 years old.
Time Frame: Baseline (week 2 or, if missing, week 3), week 24, 28 and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Score on a scale
  Week 24 - participants ≥ 10 treated with deferasirox DT (PRO): number analyzed (Participants) | 72
  Week 24 - participants ≥ 10 treated with deferasirox DT (PRO) | -0.1 (1.99)
  Week 24 - participants ≥ 10 treated with deferasirox FCT (PRO): number analyzed (Participants) | 4
  Week 24 - participants ≥ 10 treated with deferasirox FCT (PRO) | -1.0 (1.15)
  Week 28 - participants ≥ 10 treated with deferasirox DT (PRO): number analyzed (Participants) | 0
  Week 28 - participants ≥ 10 treated with deferasirox FCT (PRO): number analyzed (Participants) | 77
  Week 28 - participants ≥ 10 treated with deferasirox FCT (PRO) | 0.3 (1.84)
  Week 48 - participants ≥ 10 treated with deferasirox DT (PRO): number analyzed (Participants) | 0
  Week 48 - participants ≥ 10 treated with deferasirox FCT (PRO): number analyzed (Participants) | 75
  Week 48 - participants ≥ 10 treated with deferasirox FCT (PRO) | 0.5 (1.80)
  Week 24 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 55
  Week 24 - participants < 10 years treated with deferasirox DT (ObsRO) | -0.4 (1.33)
  Week 24 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 3
  Week 24 - participants < 10 years treated with deferasirox FCT (ObsRO) | -0.7 (1.15)
  Week 28 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 0
  Week 28 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 58
  Week 28 - participants < 10 years treated with deferasirox FCT (ObsRO) | 0.1 (2.05)
  Week 48 - participants < 10 years treated with deferasirox DT (ObsRO): number analyzed (Participants) | 0
  Week 48 - participants < 10 years treated with deferasirox FCT (ObsRO): number analyzed (Participants) | 54
  Week 48 - participants < 10 years treated with deferasirox FCT (ObsRO) | 0.1 (1.58)

11. Secondary Outcome: Change From Baseline in Gastrointestinal (GI) Symptom Score Based on GI Questionnaire
Description: The GI symptom score was calculated from responses to 5 questions of the GI questionnaire, each with a possible score of 1 to 5, for an overall possible score range of 5 to 25, where a lower score represents a less severe GI symptom and a higher score represents a more severe GI symptom.
  An observer GI symptom questionnaire was administered to those patients who were < 10 years old. The questionnaire was completed by the parents of the participants. All items and the scoring algorithm remained the same as for participants ≥ 10 years old.
Time Frame: Baseline (week -1 or, if missing, week -2), week 24, 28 and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
Score on a scale
  Week 24 - participants ≥ 10 years treated with deferasirox DT: number analyzed (Participants) | 71
  Week 24 - participants ≥ 10 years treated with deferasirox DT | 1.4 (5.53)
  Week 24 - participants ≥ 10 years treated with deferasirox FCT: number analyzed (Participants) | 4
  Week 24 - participants ≥ 10 years treated with deferasirox FCT | 5.8 (12.82)
  Week 28 - participants ≥ 10 years treated with deferasirox DT: number analyzed (Participants) | 0
  Week 28 - participants ≥ 10 years treated with deferasirox FCT: number analyzed (Participants) | 75
  Week 28 - participants ≥ 10 years treated with deferasirox FCT | -1.9 (4.33)
  Week 48 - participants ≥ 10 years treated with deferasirox DT: number analyzed (Participants) | 0
  Week 48 -participants ≥ 10 years treated with deferasirox FCT: number analyzed (Participants) | 75
  Week 48 -participants ≥ 10 years treated with deferasirox FCT | -2.2 (4.74)
  Week 24 - participants < 10 years treated with deferasirox DT: number analyzed (Participants) | 60
  Week 24 - participants < 10 years treated with deferasirox DT | 0.2 (2.78)
  Week 24 - participants < 10 years treated with deferasirox FCT: number analyzed (Participants) | 3
  Week 24 - participants < 10 years treated with deferasirox FCT | -2.0 (2.65)
  Week 28 - participants < 10 years treated with deferasirox DT: number analyzed (Participants) | 0
  Week 28 - participants < 10 years treated with deferasirox FCT: number analyzed (Participants) | 62
  Week 28 - participants < 10 years treated with deferasirox FCT | -0.5 (2.49)
  Week 48 - participants< 10 years treated with deferasirox DT: number analyzed (Participants) | 0
  Week 48 - participants < 10 years treated with deferasirox FCT: number analyzed (Participants) | 61
  Week 48 - participants < 10 years treated with deferasirox FCT | -0.6 (2.33)

12. Secondary Outcome: Change From Baseline in Serum Ferritin Levels
Description: Absolute change from baseline over time in serum ferritin levels
Time Frame: From Baseline (Day 1) up to 96 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microgram/liter (ug/L)
Arm/Group | Deferasirox DT Followed by Deferasirox FCT
Number analyzed (Participants) | 139
microgram/liter (ug/L)
  Week 2 - participants treated with deferasirox DT: number analyzed (Participants) | 108
  Week 2 - participants treated with deferasirox DT | 363.654 (323.3828)
  Week 4 - participants treated with deferasirox DT: number analyzed (Participants) | 120
  Week 4 - participants treated with deferasirox DT | 393.126 (457.8032)
  Week 8 - participants treated with deferasirox DT: number analyzed (Participants) | 121
  Week 8 - participants treated with deferasirox DT | 462.560 (427.7138)
  Week 12 - participants treated with deferasirox DT: number analyzed (Participants) | 129
  Week 12 - participants treated with deferasirox DT | 510.455 (548.6222)
  Week 16 - participants treated with deferasirox DT: number analyzed (Participants) | 131
  Week 16 - participants treated with deferasirox DT | 519.038 (508.7432)
  Week 20 - participants treated with deferasirox DT: number analyzed (Participants) | 134
  Week 20 - participants treated with deferasirox DT | 540.618 (548.2318)
  Week 24 - participants treated with deferasirox DT: number analyzed (Participants) | 130
  Week 24 - participants treated with deferasirox DT | 644.849 (629.6687)
  Week 28 - participants treated with deferasirox FCT: number analyzed (Participants) | 114
  Week 28 - participants treated with deferasirox FCT | 679.610 (701.6219)
  Week 32 - participants treated with deferasirox FCT: number analyzed (Participants) | 126
  Week 32 - participants treated with deferasirox FCT | 623.600 (629.5417)
  Week 36 - participants treated with deferasirox FCT: number analyzed (Participants) | 127
  Week 36 - participants treated with deferasirox FCT | 679.011 (674.6716)
  Week 40 - participants treated with deferasirox FCT: number analyzed (Participants) | 120
  Week 40 - participants treated with deferasirox FCT | 739.016 (659.0840)
  Week 44 - participants treated with deferasirox FCT: number analyzed (Participants) | 120
  Week 44 - participants treated with deferasirox FCT | 748.063 (647.3000)
  Week 48 - participants treated with deferasirox FCT: number analyzed (Participants) | 120
  Week 48 - participants treated with deferasirox FCT | 833.700 (788.0650)
  Week 52 - participants treated with deferasirox FCT: number analyzed (Participants) | 113
  Week 52 - participants treated with deferasirox FCT | 760.229 (798.0836)
  Week 56 - participants treated with deferasirox FCT: number analyzed (Participants) | 106
  Week 56 - participants treated with deferasirox FCT | 903.622 (832.9872)
  Week 60 - participants treated with deferasirox FCT: number analyzed (Participants) | 102
  Week 60 - participants treated with deferasirox FCT | 980.644 (994.4445)
  Week 64 - participants treated with deferasirox FCT: number analyzed (Participants) | 92
  Week 64 - participants treated with deferasirox FCT | 863.579 (854.8592)
  Week 68 - participants treated with deferasirox FCT: number analyzed (Participants) | 91
  Week 68 - participants treated with deferasirox FCT | 921.725 (860.8738)
  Week 72 - participants treated with deferasirox FCT: number analyzed (Participants) | 90
  Week 72 - participants treated with deferasirox FCT | 971.112 (872.7306)
  Week 76 - participants treated with deferasirox FCT: number analyzed (Participants) | 90
  Week 76 - participants treated with deferasirox FCT | 888.917 (869.0805)
  Week 80 - participants treated with deferasirox FCT: number analyzed (Participants) | 77
  Week 80 - participants treated with deferasirox FCT | 1005.758 (868.4338)
  Week 84 - participants treated with deferasirox FCT: number analyzed (Participants) | 87
  Week 84 - participants treated with deferasirox FCT | 1013.683 (924.5828)
  Week 88 - participants treated with deferasirox FCT: number analyzed (Participants) | 80
  Week 88 - participants treated with deferasirox FCT | 1117.849 (985.0767)
  Week 92 - participants treated with deferasirox FCT: number analyzed (Participants) | 74
  Week 92 - participants treated with deferasirox FCT | 1222.429 (1027.2565)
  Week 96 - participants treated with deferasirox FCT: number analyzed (Participants) | 74
  Week 96 - participants treated with deferasirox FCT | 1137.347 (972.1286)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs (including all-cause mortality data table) were collected from day of first dose to 30 days after last dose of study medication, assessed up to approximately 30 weeks for deferasirox DT treatment (core phase), 39 weeks for deferasirox FCT treatment (core phase) and 52 weeks for deferasirox FCT treatment (extension phase).
Description: Any sign or symptom that occurred during the study treatment plus the 30 days post treatment. Safety analyses were performed in all participants who received at least one dose of either study treatment (DT or FCT), and at least one safety assessment on or after Day 1. If, for a participant, AE start date was in deferasirox DT period and end date was in deferasirox FCT period, the participant was counted in both periods.
Groups:
- Deferasirox DT (Core Phase): Participants who were treated with deferasirox DT once daily in the core phase
- Deferasirox FCT (Core Phase): Participants who were treated with deferasirox FCT once daily in the core phase
- Deferasirox FCT (Extension Phase): Participants who were treated with deferasirox FCT once daily in the extension phase
Arm/Group | Deferasirox DT (Core Phase) | Deferasirox FCT (Core Phase) | Deferasirox FCT (Extension Phase)
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/140 | 0/116
Serious Adverse Events (participants affected / at risk) | 13/148 | 6/140 | 16/116
Other Adverse Events (participants affected / at risk) | 82/148 | 59/140 | 49/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox DT (Core Phase) (N=148) | Deferasirox FCT (Core Phase) (N=140) | Deferasirox FCT (Extension Phase) (N=116)
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Optic nerve cupping (Eye disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 2
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Ecthyma (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox DT (Core Phase) (N=148) | Deferasirox FCT (Core Phase) (N=140) | Deferasirox FCT (Extension Phase) (N=116)
Diarrhoea (Gastrointestinal disorders) | 16 | 5 | 2
Pyrexia (General disorders) | 7 | 8 | 5
Hepatomegaly (Hepatobiliary disorders) | 8 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 7 | 3
Pharyngitis (Infections and infestations) | 7 | 6 | 6
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 4
Urinary tract infection (Infections and infestations) | 9 | 3 | 3
Serum ferritin increased (Investigations) | 8 | 2 | 1
Urine protein/creatinine ratio increased (Investigations) | 13 | 12 | 7
Proteinuria (Renal and urinary disorders) | 8 | 9 | 12
Hepatic enzyme increased (Investigations) | 5 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT02993224/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT02993224/SAP_001.pdf